CLINICAL TRIAL: NCT03823105
Title: Validation of Non-invasive Miniature Optical Sensors for Scoring Sleep Stages: a Prospective, Method-comparison, Proof of Concept, Single-centre Phase IV Study
Brief Title: Validation of Non-invasive Miniature Optical Sensors for Scoring Sleep Stages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-00917
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Sleep-Wake Disorders; Healthy
Keywords: Sleep apnea; Hypersomnia; Parasomnia
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes; Disorders of Excessive Somnolence; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nocturnal Recording (Experimental): Recording of photoplethysmographic pulse wave and accelerometry with two devices (OHR Tracker, PulseWatch) in parallel to the standard polysomnography
  Interventions: Device: OHR Tracker and PulseWatch

INTERVENTIONS:
Device: OHR Tracker and PulseWatch — Category A (ClinO). Medical study with CE-marked medical devices to photoplethysmographic measure heart rate, heart rate variability, and pulse wave and accelerometric data

SUMMARY:
Validation of two devices with optical sensor in healthy participants and patients with sleep wake disorders.

DETAILED DESCRIPTION:
The objective of this study is to evaluate and optimize a method of detecting sleep and sleep stages based on a new algorithm combining actigraphy and heart rate variability (measured by optical analysis of the pulse wave) to determine sleep architecture (segmented into three phases: WAKE, REM and NREM) with high accuracy compared to the gold standard polysomnography.

ELIGIBILITY:
Patients with sleep wake disorders

Inclusion Criteria:

* 18 ≤ Age ≤ 80 years
* Suspected sleep wake disorder (sleep apnea, sleep movement disorders, hypersomnia, parasomnia)
* Written informed consent

Exclusion Criteria:

* Skin condition with eczema or damaged skin
* Ischemia (cutaneous)
* Allergy against nickel
* Allergy against silicone
* Current treatment with vasoactive drugs (e.g. beta-blockers, calcium channel antagonists, nitroglycerin, etc.) and/or antidepressive drugs (e.g. serotonin reuptake inhibitors, etc.).
* Known infection with multiresistant bacteria
* Implanted devices (e.g. pacemaker, pumps)
* Rhythmogenic heart disease (e.g. resting heart rate > 120/min)
* Severe or untreated arterial hypertension (blood pressure > 140mmHg systolic, >90mmHg diastolic)
* Hypotension (blood pressure < 90mmHg systolic, < 60 mmHg diastolic)
* Current alcohol or drug abuse, alcohol consumption the same day as the study
* Consumption of coffee 7h before
* Dark skin pigmentation
* Severe metabolic disease (e.g. diabetes)
* Pregnancy or lactation
* Physical handicap effecting the two arms
* Wound in the wrist region
* Too large or too small wrist

Healthy subjects

Inclusion criteria:

* 18 ≤ Age ≤ 80 years
* Written informed consent

Exclusion criteria:

* Skin condition with eczema or damaged skin
* Ischemia (cutaneous)
* Allergy against nickel
* Allergy against silicone
* Any Medication (except birth control pill)
* Known infection with multiresistant bacteria
* Implanted devices (e.g. pacemaker, pumps)
* Rhythmogenic heart disease (e.g. resting heart rate > 120/min)
* Severe or untreated arterial hypertension (blood pressure > 140mmHg systolic, >90mmHg diastolic)
* Hypotension (blood pressure < 90mmHg systolic, < 60 mmHg diastolic)
* Current alcohol or drug abuse, alcohol consumption the same day as the study
* Consumption of coffee 7h before
* Implanted devices (e.g. pacemaker, pumps)
* Known sleep-wake disorders
* Dark skin pigmentation
* Severe metabolic disease (e.g. diabetes)
* Pregnancy or lactation
* Physical handicap effecting the two arms
* Wound in the wrist region
* Too large or too small wrist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST) and sleep architecture (distribution of sleep stages) | 1 night
  Diagnostic accuracy of the new algorithm compared to the Gold Standard full polysomnography
The total time in non-REM sleep (stages 1-3), REM sleep, and awake after sleep onset | 1 night
  Diagnostic accuracy of the new algorithm compared to the Gold Standard full polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian R. Ott, MD, Principal Investigator — University Hospital Berne, Department of Pulmonary Medicine
Locations (1):
- University Hospital Bern (Inselspital), Department of Pulmonary Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided